CLINICAL TRIAL: NCT03231098
Title: A Quantitative and Comparative Study for the Detection of Group A β-Hemolytic Streptococci in Patient Throat Gargle
Brief Title: Detection of GABHS in Throat Gargle
Status: Completed | Type: Observational
Sponsor: Gargle Tech (Industry)
Responsible Party: Sponsor
Other Study IDs: STRP.P001
Record Dates: First submitted 2017-07-23; First posted 2017-07-27 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Group A Streptococcus: B Hemolytic Pharyngitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The objective of this study is to investigate the use of patient throat gargle as an alternative to throat swabbing for the diagnosis of pharyngitis caused by Group A β-Hemolytic Streptococcus (GABHS) infection, also known as strep throat.

DETAILED DESCRIPTION:
The aim of this study is to procure a detailed quantitative and qualitative analysis of GABHS present in patient throat gargle and to compare various culturing techniques and immunoassay methods for efficient and effective GABHS detection from gargle fluid. During the course of this clinical trial, the following specimen samples will be collected from each participating patient: the patient will first be asked to gargle 10-15 mL of sterile saline to obtain a gargle sample, and then the patient will be subjected to two routine standard throat swabs. These specimen samples will be properly discarded after processing and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Suspected of suffering from GABHS pharyngitis.
* Able to communicate with study personnel (English or Hebrew).
* Able to understand oral and written information about the study.
* Willing to provide written informed consent to participate in the study.

Exclusion Criteria:

* Not capable of gargling 10-15 mL fluid.
* Diagnosed or self-reported pregnancy.
* History of dementia, cognitive impairment, or psychiatric or mental disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients age 18 years and older who present to the study site with complaints of sore throat and are suspected of suffering from GABHS pharyngitis.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-02-16 (Actual)

PRIMARY OUTCOMES:
Comparative: Method sensitivity to investigate method effectiveness. | Through study completion, about 9 months
  Compare sensitivity of each gargle fluid GABHS detection method.
Comparative: Method specificity to investigate method effectiveness. | Through study completion, about 9 months
  Compare specificity of each gargle fluid GABHS detection method.

SECONDARY OUTCOMES:
Quantitative: Average GABHS in gargle. | Through study completion, about 9 months
  Average number of total GABHS bacteria collected in throat gargle samples.
Quantitative: Minimum GABHS in gargle. | Through study completion, about 9 months
  Minimum number of total GABHS bacteria collected in throat gargle samples.

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Alpert, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- TEREM Ha'Gdud Ha'Ivri Family Clinic, Jerusalem, Israel

REFERENCES:
- [Background] Karabay O, Ekerbicer H, Yilmaz F. Efficacy of throat gargling for detection of group a beta-hemolytic streptococcus. Jpn J Infect Dis. 2005 Feb;58(1):39-40. PMID 15728991